CLINICAL TRIAL: NCT06519123
Title: Assessing the Impact of Ambient Digital Scribes Populating Clinical Notes on Patient and Clinician Satisfaction
Brief Title: Ambient Digital Scribes Populating Clinical Notes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00116295
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-09

CONDITIONS: Patient Satisfaction; Clinician Satisfaction
Keywords: Ambient Digital Scribes; AI; Communication
MeSH Terms: conditions — Patient Satisfaction; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population - Clinicians and Patients (Experimental): Clinicians will audio record 4 patient encounters on two separate days each (240 encounters).
  Interventions: Other: Ambient Digital Scribes

INTERVENTIONS:
Other: Ambient Digital Scribes — AI technology used to populate clinical notes.

SUMMARY:
The purpose of this study is to assess the impact of Ambient Digital Scribes that will automatically record clinical encounters and use AI technology to populate clinical notes. The investigators expect that when clinicians do not need to either write notes during the clinical encounter and can instead face patients when talking, several effects could result, including 1) patients report higher satisfaction with the visit 2) clinicians report less burnout, and 3) clinician-patient communication includes more evidence-based tools that indicate high quality communication.

DETAILED DESCRIPTION:
Effective communication forms the foundation of high-quality care. Communication includes verbal and nonverbal channels, with nonverbal communication playing a large role in acknowledging and responding to patient concerns. Effective communication has been negatively affected by the introduction of the electronic health record and required documentation. Clinicians often attend to the computer, writing notes during the encounter, which can lead to missing emotional cues from patients. Missing this key information can leave patients feeling dismissed, not heard, and can lead to lower comprehension and adherence. Further, the amount clinicians need to document often cannot occur solely in the encounter, leading to clinicians working after hours to finish their notes. The cumulative effect of the change in communication and required documentation has been a strong predictor of burnout among clinicians.

The introduction of AI into healthcare might have a positive impact on both efficiency and communication, thus resulting in higher clinician and patient satisfaction. With the advent of Ambient Digital Scribes and AI potentially populating notes, clinicians can have the opportunity to attend fully to patients both verbally and nonverbally. Patients likely will feel more heard, valued, and can ask questions, leading to higher comprehension and adherence. Clinicians might feel the burden of documentation lifted, might be more efficient, and feel more satisfied by providing the care they desire.

To test the impact of Ambient Digital Scribes, the investigators propose a sub-study to the approved project (Pro00115827) where the investigators will audio record clinicians in usual care before they are assigned to the two different scribing programs. The investigators will assess patient outcomes, namely perceived empathy and patient satisfaction, and clinician burnout. The investigators also will code audio recorded encounters to assess: 1) reflective statements (showing active listening), 2) empathic responses to empathic opportunities, 3) patient question-asking, and 4) length of encounter.

ELIGIBILITY:
Patient Inclusion Criteria:

* 18 years or older
* able to speak and read English

Patient Exclusion Criteria:

* unable to speak and read English

Clinician Inclusion Criteria:

* delivering care in a clinic in which Ambient Digital Scribes are being employed

Clinician Exclusion Criteria:

* not delivering care in a clinic in which Ambient Digital Scribes are being employed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Patient-perceived clinician empathy | through study completion, an average of 2 months
  Patient perceived empathy will be assessed via post doctor appointment administered survey.
Patient Satisfaction | through study completion, an average of 2 months
  Patient satisfaction will be assessed via post doctor appointment administered survey.

SECONDARY OUTCOMES:
Clinician Satisfaction as measured by level of burnout | through study completion, an average of 2 months
  Assessed by clinician-reported levels of burnout via survey.
Clinician Communication | through study completion, an average of 2 months
  Communication will be coded for reflective statements (showing active listening), empathic responses to empathic opportunities, patient question-asking, and length of encounter.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No